CLINICAL TRIAL: NCT04279925
Title: A Clinical Trial of Locally Made Titanium Miniplate and Screw in Maxillofacial Fractures Management
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Aerosol risk of COVID-19 spread resulting a slow subject recruitment
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Prasetyanugraheni Kreshanti, SpBP-RE (KKF), Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1085/UN2.F1/ETIK/PPM.0002/2019
Record Dates: First submitted 2020-02-10; First posted 2020-02-21 (Actual); Results first posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Maxillofacial Injuries; Maxillofacial Prosthesis Implantation; Fracture Fixation, Internal
MeSH Terms: conditions — Maxillofacial Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: a radiologist consultant as a blinded independent evaluator will assess the bone density score in each subject.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Locally-made Miniplate and screw (Experimental): Locally-made miniplate and screw produced by the Faculty of Engineering Universitas Indonesia.
  Interventions: Device: ORIF (Open reduction internal fixation): locally-made miniplate and screw
- Imported Miniplate and screw (Active Comparator): Biomet® miniplate 1.5 and screw 1.5 produced by Biomet, included in the Lorenz® Plating System Midface.
  Interventions: Device: ORIF: Imported miniplate and screw

INTERVENTIONS:
Device: ORIF (Open reduction internal fixation): locally-made miniplate and screw — Fracture lines in this group underwent open reduction internal fixation (ORIF) procedure which consists of realignment of the bone achieved from surgical mean and stabilization of the bone fragments by using locally-made miniplate and screw produced by the Faculty of Engineering Universitas Indonesia. The plate used in the study is a straight plate with 4 and 5 holes with the dimension of 17mm long, 4 mm wide and 0.56 mm thick.
  Arms: Locally-made Miniplate and screw
Device: ORIF: Imported miniplate and screw — Fracture lines in this group underwent open reduction internal fixation (ORIF) procedure which consists of realignment of the bone achieved from surgical mean and stabilization of the bone fragments by using Biomet® miniplate 1.5 produced by Biomet, included in the Lorenz® Plating System Midface. The particular plate used in the study is a straight plate with 4 holes, 17mm length and 0.6mm thick, coded 01-7047 in the catalog. Biomet® screw 1.5 utilized in this study is also produced by Biomet, included in the Lorenz® Plating System Midface. The dimension of the screw is 4mm length, 1.5 mm diameter, and coded 91-6104 1.5 mm X-Drive Self drilling screws.
  Arms: Imported Miniplate and screw

SUMMARY:
The study is a blind randomized clinical study on patients with midface maxillofacial fractures coming to Cipto Mangunkusumo Hospital. The subject is the fracture line who met the inclusion criteria and randomly allocated into the study (locally-made miniplate and screw) and control (BIOMET® miniplate and screw) group through a predetermined randomization list. The healing process is follow up using non-contrast head computed tomography immediately after surgery as a baseline, and 3 months post-op. Afterward, a radiologist consultant as a blinded evaluator will evaluate the score of bone density, and screw loosening, while local tissue reaction after fixation evaluates during the patient's visit outpatient clinic. All scores from points of the evaluation group will be collected and going to statistically evaluated using independent t-test or Mann Whitney test depending on the distribution of the data

ELIGIBILITY:
Inclusion Criteria:

* Midface fracture with the indication of surgery
* Midface fracture sustained within 2 weeks

Exclusion Criteria:

* Comminuted and defect fracture
* Midface fracture on patients with systemic diseases affecting bone healing.
* Midface fracture in children
* Midface fracture in multiple trauma patients with neurological deterioration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto mangunkusumo National Hospital, Jakarta Pusat, Central, Indonesia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: * participants signed the informed consent form and declare that they want to be enrolled as subjects and obey all the instructions given postoperatively
  * They were showered with chlorhexidine 4% soap one day before surgery
Period: Overall Study
Arm/Group | Locally-made Miniplate and Screw | Imported Miniplate and Screw
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Locally-made Miniplate and Screw | Imported Miniplate and Screw | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 5 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 5 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Indonesia | 4 | 5 | 9
Bone density [Mean (Standard Deviation); unit: Hounsfield Unit (HU)] — The Hounsfield unit (HU) is a relative quantitative measurement of radio density used by radiologists in the interpretation of computed tomography (CT) images.The Hounsfield unit, also referred to as the CT unit, is then calculated based on a linear transformation of the baseline linear attenuation coefficient of the X-ray beam, where air is usually -1000 HU and air 0 HU. The HU for bones ranges from 148 (cancellous bones) to 3000 (dense bones), -700 to 225 HU for soft tissues, -205 to -72 HU for fat, and -5 to 139 for muscle.
  Hounsfield Unit (HU) | 111.3080 (182.8720) | 251.2050 (214.5910) | 181.2565 (198.7315)

OUTCOME MEASURES:

1. Primary Outcome: Bone Density
Description: The Hounsfield unit (HU) is a relative quantitative measurement of radio density used by radiologists in the interpretation of computed tomography (CT) images.The Hounsfield unit, also referred to as the CT unit, is then calculated based on a linear transformation of the baseline linear attenuation coefficient of the X-ray beam, where air is usually -1000 HU and air 0 HU. The HU for bones ranges from 148 (cancellous bones) to 3000 (dense bones), -700 to 225 HU for soft tissues, -205 to -72 HU for fat, and -5 to 139 for muscle.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: Hounsfield Unit (HU)
Groups:
- Locally-made Miniplate and Screw: Fracture lines in this group underwent open reduction internal fixation (ORIF) procedure which consists of realignment of the bone achieved from surgical mean and stabilization of the bone fragments by using locally-made miniplate and screw produced by the Faculty of Engineering Universitas Indonesia. The plate used in the study is a straight plate with 4 and 5 holes with the dimension of 17mm long, 4 mm wide and 0.56 mm thick.
- Imported Miniplate and Screw: Fracture lines in this group underwent open reduction internal fixation (ORIF) procedure which consists of realignment of the bone achieved from surgical mean and stabilization of the bone fragments by using Biomet® miniplate 1.5 produced by Biomet, included in the Lorenz® Plating System Midface. The particular plate used in the study is a straight plate with 4 holes, 17mm length and 0.6mm thick, coded 01-7047 in the catalog. Biomet® screw 1.5 utilized in this study is also produced by Biomet, included in the Lorenz® Plating System Midface. The dimension of the screw is 4mm length, 1.5 mm diameter, and coded 91-6104 1.5 mm X-Drive Self drilling screws.
Arm/Group | Locally-made Miniplate and Screw | Imported Miniplate and Screw
Number analyzed (Participants) | 4 | 5
Hounsfield Unit (HU) | 111.3080 [-90.2572 to 592.6672] | 251.2050 [-115.758 to 338.3736]

2. Secondary Outcome: Screw Loosening (Yes/No)
Description: Screw loosening will be recorded, whether it is present or not. It will be evaluated by a radiologist consultant after the subject completed all their Head CT evaluation. The outcome will be presented as the percentage of patients with screw loosening, evaluated from head CT Scan.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Locally-made Miniplate and Screw | Imported Miniplate and Screw
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

3. Secondary Outcome: Tissue Reaction (Yes/No)
Description: Clinical signs of local inflammation process, will be recorded by the end of the 3rd week during patient's visit in outpatient clinic. It will be evaluated by consultants of craniomaxillofacial surgery. The outcome will be presented as the number of patients with signs of local inflammation.
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Locally-made Miniplate and Screw | Imported Miniplate and Screw
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Locally-made Miniplate and Screw | Imported Miniplate and Screw
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, it is difficult to reach the number of samples as planned, the clinical study was underpowered. The clinical study will be extended (currently submitting amendment of ethical clearance), to reach more power in the study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT04279925/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT04279925/ICF_001.pdf